CLINICAL TRIAL: NCT01238146
Title: A Phase I/II Trial of Rituximab, Bendamustine, and Obatoclax in Patients With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma
Brief Title: Obatoclax Mesylate, Rituximab, and Bendamustine Hydrochloride in Treating Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No patients accrued.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02536; OSU-10040; U01CA076576 (NIH); CDR0000687197 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Splenic Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; obatoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive obatoclax mesylate IV over 3 hours on days 1-3, rituximab IV over 4-8 hours on day 1, and bendamustine hydrochloride IV over 30 minutes on days 1-2.
  Interventions: Drug: bendamustine hydrochloride; Drug: obatoclax mesylate; Biological: rituximab
- Arm II (Experimental): Patients receive rituximab and bendamustine hydrochloride as in arm I.
  Interventions: Drug: bendamustine hydrochloride; Biological: rituximab

INTERVENTIONS:
Drug: bendamustine hydrochloride — Given IV
  Other Names: bendamustin hydrochloride; bendamustine; cytostasan hydrochloride; Treanda
Drug: obatoclax mesylate — Given IV
  Other Names: GX15-070MS
  Arms: Arm I
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan

SUMMARY:
This phase I/II trial is studying the side effects and the best dose of obatoclax mesylate when given together with rituximab and bendamustine hydrochloride to see how well it works compared with rituximab and bendamustine hydrochloride alone in treating patients with relapsed or refractory non-Hodgkin lymphoma. Obatoclax mesylate may stop the growth of cancer cells by blocking some of the proteins needed for cell growth. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and help kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as bendamustine hydrochloride, also work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving obatoclax mesylate together with rituximab and bendamustine hydrochloride may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose-limiting toxicity (DLT) and maximum-tolerated dose (MTD) of the combination of obatoclax mesylate, rituximab, and bendamustine hydrochloride in patients with relapsed or refractory, indolent, B-cell non-Hodgkin lymphoma (phase I).

II. To define the qualitative and quantitative toxicities of the combination of obatoclax mesylate, rituximab, and bendamustine (phase I).

III. To detect an improvement in median progression-free survival (PFS) from 6 to 12 months with the addition of obatoclax mesylate to rituximab and bendamustine hydrochloride in patients with indolent B-cell non-Hodgkin lymphoma (phase II).

SECONDARY OBJECTIVES:

I. To determine the overall objective response rate to the combination of obatoclax mesylate, rituximab, and bendamustine versus rituximab and bendamustine hydrochloride in patients with relapsed or refractory, indolent, B-cell non-Hodgkin lymphoma.

II. To characterize two-year PFS of patients with indolent B-cell non-Hodgkin lymphoma receiving obatoclax mesylate, rituximab, and bendamustine hydrochloride versus rituximab and bendamustine hydrochloride.

III. To assess the pharmacokinetics of obatoclax mesylate in patients with relapsed or refractory, indolent, B-cell non-Hodgkin lymphoma.

IV. To assess the pharmacokinetics of the combination of bendamustine hydrochloride and obatoclax mesylate in patients with relapsed or refractory, indolent, B-cell non-Hodgkin lymphoma.

V. To determine the effects of the combination of rituximab, bendamustine hydrochloride, and obatoclax mesylate on histone-oligodeoxynucleotide (ODNA) and levels of activated Bax and Bak pro-apoptotic proteins in peripheral blood mononuclear cells and bone marrow aspirate specimens.

VI. To identify associations of genetic polymorphisms in drug-metabolizing enzymes, transporters, or target genes with pharmacokinetics, pharmacodynamics, or clinical outcomes.

OUTLINE: This is a phase I, dose-escalation study of obatoclax mesylate followed by a randomized phase II study.

PHASE I: Patients receive obatoclax mesylate IV over 3 hours on days 1-3, rituximab IV over 4-8 hours on day 1 (day 3 of course 1), and bendamustine hydrochloride IV over 30 minutes on day 1-2 (day 2-3 of course 1). Treatment repeats every 28 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are stratified according to prior bendamustine hydrochloride (yes vs no). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive obatoclax mesylate IV over 3 hours on days 1-3, rituximab IV over 4-8 hours on day 1, and bendamustine hydrochloride IV over 30 minutes on days 1-2.

ARM II: Patients receive rituximab and bendamustine hydrochloride as in arm I.

In both arms, treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood and bone marrow sample collection at baseline and periodically during study for pharmacokinetics, pharmacodynamic, and pharmacogenetic studies.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed indolent B-cell non-Hodgkin lymphoma (NHL), including any of the following subtypes recognized by WHO classification:

  * Marginal zone lymphoma
  * Lymphoplasmacytic lymphoma
  * Follicular lymphoma
  * Mantle cell lymphoma
* Transformed lymphoma from a low-grade, indolent NHL allowed provided patient has received ≥ 1 prior therapy for indolent disease
* Must have received ≥ 1 prior therapy
* Relapsed disease after autologous or allogeneic stem cell transplantation (SCT) allowed (phase I)

  * No relapse after allogeneic SCT (phase II)
* No known CNS lymphoma
* ECOG performance status 0-2
* ANC ≥ 1,000/µL
* Platelet count ≥ 50,000/µL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception prior to and for the duration of study participation
* No active hepatitis B infection

  * Patients with a history of hepatitis B (surface antigen or core antibody positive) must take lamivudine or equivalent during study therapy
* No history of documented human anti-globulin antibodies, or a history of allergic reactions attributed to compounds of similar chemical or biologic composition to rituximab, bendamustine hydrochloride, or obatoclax mesylate
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness and/or social situations that would limit compliance with study requirements
* HIV infection allowed provided patient meets the following criteria:

  * No evidence of co-infection with hepatitis B or C
  * CD4 cell count ≥ 400/mm³
  * No evidence of resistant strains of HIV
  * HIV viral load ≤ 10,000 copies HIV RNA/mL for patients not on anti-HIV combination antiretroviral therapy OR HIV viral load ≤ 50,000 copies HIV RNA/mL for patients on anti-HIV therapy
  * No history of AIDS-defining conditions
* No active secondary malignancy except for non-melanomatous skin cancer
* No other concurrent investigational agents
* Prior bendamustine hydrochloride allowed provided patient has completed a bendamustine-containing regimen within the past 6 months and achieved a partial response or better
* More than 4 weeks since prior chemotherapy or radiotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerable dose, defined as the dose level beneath which 2 or more of 6 patients experience DLT (phase I) | 28 days
  Graded using CTCAE version 4 criteria. DLTs are defined as grade 3-4 neutropenia or thrombocytopenia that persists beyond day 42; grade 4 febrile neutropenia or infection; grade 3 febrile neutropenia or infection that fails to resolve within 7days, grade 3-4 somnolence, ataxia, or confusion that requires inpatient admission on day 1 for observation and prevents patient discharge from outpatient clinic, or other grade 3-4 non-hematologic toxicity excluding infection.
Change in median progression-free survival (PFS) (phase II) | From 6 to 12 months
  Estimated using the method of Kaplan-Meier.

SECONDARY OUTCOMES:
Overall objective response rate (phase II) | Up to 3 years
  95% confidence intervals will be provided.
PFS (phase II) | From the date of start of therapy to disease progression or death, whichever occurs first, assessed at 2 years
  Estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Christian, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States